CLINICAL TRIAL: NCT04519190
Title: Screening for Atrial Fibrillation With Prolonged Continuous Single-lead ECG Devices in High-risk Patients
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Huashan Hospital (Other)
Responsible Party: Principal Investigator, Xiufang Gao, Associate chief physian, Huashan Hospital
Other Study IDs: SAFE-high risk
Record Dates: First submitted 2020-08-15; First posted 2020-08-19 (Actual); Last update posted 2020-08-19 (Actual); Status verified 2020-08

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Prolonged continuous single-lead ECG monitor — We use Smartpatch, a listed ambulatory electrocardiographic system that can continuously record and save patients' cardiac rhythm for up to 45 days.
Diagnostic Test: Intermittent ECG monitor — When using Smartpatch, we can set time markers by pressing the button on the device. We ask our subjects to press that button twice a day and also when they feel any discomfort. Analyzing the ECG 1 minute after those time markers can serve as a surrogate for intermittent ECG monitor.
Diagnostic Test: Routine practice — Perform pulse palpation and also ECG if irregular rhythm is found.

SUMMARY:
Atrial fibrillation(AF) can be asymptomatic and thus left unidentified in many people, but holds potential risk of lethal complications such as stroke and congestive heart failure. With different screening strategy, the screening result will be different. The longer the monitoring period is, the higher chances AF episodes can be identified, but with greater cost and lower compliance. Therefore, in this study, the investigators want to find the most cost-effective method for AF screening in high risk population with prolonged continuous single-lead ECG device.

ELIGIBILITY:
We created a score system as to predict AF risk.

1. Age ≥ 75: 2points Age between 65-74: 1point
2. Male: 1point
3. Stroke: Typical symptoms of acute stroke with multiple foci on imaging examination: 5points Typical symptoms of acute stroke with single or uncertain lesion on imaging: 3 points Imaging examination shows old cerebral infarction, transient ischemic attack(TIA), lacunar infarction with clear symptoms: 2points
4. Congestive heart failure: Ejection fraction(EF)≥50%, N terminal pro-brain natriuretic peptide(NT pro-BNP)>1500 pg/mL: 1point EF 40-49%: 2points EF<40%: 4points
5. Echocardiography: Mitral stenosis or regurgitation, aortic stenosis or regurgitation: moderate degree and above: 2points Left atrial anterior-posterior diameter: 40-49mm: 1point Left atrial anterior-posterior diameter: ≥50mm: 2points
6. Vascular disease: History of myocardial infarction, percutaneous coronary intervention(PCI) or coronary artery bypass graft(CABG): 2points Clear history of peripheral arterial obstruction: 3points
7. Hypertension: Blood pressure controlled: 1point Blood pressure uncontrolled(Systolic blood pressure>160mmHg): 2points
8. Diabetic mellitus: Plasma glucose level controlled:1point Plasma glucose level uncontrolled(HBA1c>7):2points i:Chronic kidney disease: estimated glomerular filtration rate(eGFR) 30-49: 1point eGFR <30: 2points j:Sleep apnea syndrome: 1point k:Chronic obstructive pulmonary disease: 1point l:Thyroid disease: 1point

Inclusion Criteria:

* 1.Age between 18-85 2.Score ≥5points in the above scoring system 3.Volunteer to participate in the study

Exclusion Criteria:

* 1.Clear history of atrial flutter or atrial fibrillation 2.History of pacemaker implacement 3.Already on anticoagulation therapy 4.History of severe contact dermatitis 5.ECG recorded by our device unrecognizable 6.Patients with end-stage disease or at advanced stage of cancer with life expectancy less than 1 year

Ages: 18 Years to 85 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Subjects who holds several risk factors for AF but not yet diagnosed.
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2020-08-25 (Estimated); Primary Completion 2023-08-31 (Estimated); Study Completion 2023-08-31 (Estimated)

PRIMARY OUTCOMES:
Number of participates with AF episodes identified using continuous ECG monitoring compared to routine practice. | 2020-2023
  Some atrial fibrillation patients may be left undiagnosed by routine practice due to several reasons. On ECG, AF episodes are defined as irregularly irregular QRS complex with disappearance of P wave that last over 30 seconds. A routine ECG examination may not able to capture AF episodes, however, by monitoring the subjects' cardiac rhythm continuously for a prolonged time period, we can detect asymptomatic AF episodes with higher sensitivity that would have been missed. And by further analyzing the detection rates of different monitoring periods, we can find out the most cost-effective monitoring duration and pattern.